CLINICAL TRIAL: NCT05323435
Title: A Multicenter, Randomized, Observer-Blinded, Active-Controlled Phase II Study to Evaluate the Immunogenicity and Safety of One Dose Booster by Recombinant Two-Component COVID-19 Vaccine (CHO Cell) in Adults Aged 18 Years and Older
Brief Title: Immunogenicity and Safety Study of Recombinant Two-Component COVID-19 Vaccine (CHO Cell)(ReCOV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Rec-Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REC611C302
Record Dates: First submitted 2022-04-11; First posted 2022-04-12 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Recombinant Two-Component COVID-19 Vaccine (CHO cell), 20μg (Experimental): Antigen: NTD-RBD-foldon protein, sodium dihydrogen phosphate, disodium hydrogen phosphate, sucrose, glycine, polysorbate 80 Adjuvant (BFA03): squalene, alpha-tocopherol, polysorbate 80, sodium chloride, potassium chloride, disodium hydrogen phosphate, potassium dihydrogen phosphate (ReCOV for short, 20μg)
  Interventions: Biological: Recombinant two-component COVID-19 vaccine (CHO cell)
- Recombinant Two-Component COVID-19 Vaccine (CHO cell), 40μg (Experimental): Antigen: NTD-RBD-foldon protein, sodium dihydrogen phosphate, disodium hydrogen phosphate, sucrose, glycine, polysorbate 80 Adjuvant (BFA03): squalene, alpha-tocopherol, polysorbate 80, sodium chloride, potassium chloride, disodium hydrogen phosphate, potassium dihydrogen phosphate (ReCOV for short, 40μg)
  Interventions: Biological: Recombinant two-component COVID-19 vaccine (CHO cell)
- COVID-19 Vaccine (Vero Cell), Inactivated (Active Comparator): Antigen: inactivated SARS-CoV-2 Virus (19nCoV-CDC-Tan-HB02 strain) Adjuvant: aluminum hydroxide Excipients: disodium hydrogen phosphate, sodium dihydrogen phosphate, sodium chloride
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated

INTERVENTIONS:
Biological: Recombinant two-component COVID-19 vaccine (CHO cell) — Before reconstitution: Lyophilized powder for reconstitution in single-use vials After reconstitution with BFA03 adjuvant: Milk-white solution with no visible foreign matter
  Other Names: ReCOV
  Arms: Recombinant Two-Component COVID-19 Vaccine (CHO cell), 20μg; Recombinant Two-Component COVID-19 Vaccine (CHO cell), 40μg
Biological: COVID-19 Vaccine (Vero Cell), Inactivated — Milky-white suspension.Stratified precipitate may form which can be dispersed by shaking
  Arms: COVID-19 Vaccine (Vero Cell), Inactivated

SUMMARY:
This is a multicenter, randomized, observer-blinded, active-controlled Phase II study to evaluate the immunogenicity, safety and reactogenicity of the low dose (20μg) and high dose (40μg) of ReCOV, when administered as a booster to healthy adults aged 18 to 65 years who have completed two or three doses vaccination (prioritized two doses). Estimate 300 participants.

DETAILED DESCRIPTION:
The study is a multicenter, randomized, observer-blinded, active-controlled trial. About 300 eligible participants will be randomized equally (1:1:1) into 20 μg ReCOV group, 40 μg ReCOV group, and the control vaccine [COVID-19 Vaccine (Vero Cell), Inactivated] group, respectively, stratified by age (18 to < 50 years, ≥ 50 to ≤ 65 years) and the duration since the last dose of primary vaccination (90~180 days, 181~365 days).

All Participants will be observed for 30 minutes after study vaccination at study site if Participants will be asked to record solicited AEs within 7 days and unsolicited AEs within28 days. After 28 days post the study vaccination，all participants will have 2 on-site safety follow-up Visits on Day 90 (±15days) and on Day 180 (±15days) after the study vaccination to collect serious adverse evens (SAEs), adverse events of special interest (AESIs). During the study period, they can spontaneously report any adverse events (AEs) they experienced at any time.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 65 years (included).
2. Able and willing to comply with all study requirements.
3. Willing to allow the investigators to discuss the volunteers' medical history with his/her general practitioner/personal doctors and access all medical records which are relevant to study procedures.
4. Healthy adults, or adults with stable medical condition who have a pre-existing medical condition that does not meet any exclusion criteria. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrollment.
5. Have completed two doses vaccination by inactivated COVID-19 vaccine prior to the study vaccination. The duration since the last primary vaccination is 90~365 days (included) for both Phase II and Phase III stages.
6. For females of childbearing potential only, willing to practice continuous effective contraception till 90 days after the study vaccination, and have negative pregnancy tests before study vaccination.

   * Nonchildbearing potential is defined as surgically sterile (history of bilateral tubal ligation, bilateral oophorectomy, hysterectomy) or postmenopausal (defined as amenorrhea for ≥ 12 consecutive months prior to Screening without an alternative medical cause). A follicle-stimulating hormone (FSH) level may be measured at the discretion of investigator to confirm postmenopausal status.
   * The effective contraceptive methods include sexual abstinence or adequate contraceptive measures such as intrauterine or implanted contraceptive device, oral contraceptives, injected or implanted contraceptives, sustained-release topical contraceptives, condoms (male), diaphragm, and cervical cap, etc.
7. Males participating in this study who are involved in heterosexual activity must agree to practice adequate contraception (as described above) and refrain from donating sperm till 90 days after receiving the study vaccination.
8. Agreement to refrain from blood donation during the study.
9. Provide written informed consent form (ICF) prior to study enrollment.

Exclusion Criteria:

1. Laboratory confirmed SARS-CoV-2 infection, defined by the result of SARS-CoV-2 RT-PCR assay is positive.
2. Medical history of COVID-19 disease with confirmed clinical diagnosis.
3. Fever (oral temperature ≥ 37.5°C / axillary temperature ≥ 37.3°C) on the day of vaccination. Or having fever within recent 72 hours before the vaccination.
4. Having abnormal results of clinical laboratory testing during screening, which is judged by the investigator with clinical significance, including the hematology, liver function, renal function, other blood chemistry, and coagulation function.
5. History of severe allergic disease or reactions likely to be exacerbated by any component of ReCOV or COVID-19 Vaccine (Vero Cell), Inactivated, such as allergic shock, allergic laryngeal edema, allergic purpura, thrombocytopaenic purpura, local hypersensitive necrosis reaction (Arthus reaction), prior history of serious adverse reaction to any vaccine or drug, such as allergy, urticaria eczema, dyspnea, and angioneurotic edema.
6. Having malignant tumor (except for skin basal cell carcinoma or carcinoma uterine cervix in situ), immune disease (e.g., human immunodeficiency virus [HIV] infection, systemic lupus erythematosus, rheumatoid arthritis, alienia or splenectomy, and other immune disease that may influence immune response at the investigator's discretion).
7. Having severe and/or uncontrolled conditions, including but not limited to, acute infectious disease, cardiovascular disease, respiratory disease (including tuberculosis under anti-tuberculosis therapy), gastrointestinal disease, liver disease, renal disease, hematology disease, endocrine disorder, psychiatric condition and neurological illness (e.g., medical or family history of seizure, epilepsy, encephalopathy). Mild/moderate well-controlled comorbidities are allowed to participate.
8. Having bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following intramuscular injections or venipuncture.
9. Received immunosuppressant or other immunomodulators, antiallergic therapy, or cytotoxicity therapy for 14 or more consecutive days within 6 months before the study vaccination. Local administration of immunosuppressant or immunomodulator is allowed (e.g., ointment, eye drops, inhalation, or nasal spray). Drugs for local administration should not be given at a dose over the recommended level in package insert or participants should have no signs of systemic exposure.
10. Administration of immunoglobulin and/or blood product within 3 months before the study vaccination or plan to use that during the study.
11. Continuous use of anticoagulants, such as coumarins and related anticoagulants (e.g., warfarin) or novel oral anticoagulants (e.g., apixaban, rivaroxaban, dabigatran and edoxaban).
12. Used other investigational drug or interventional device within 1 month before the study vaccination or plan to use that during the study, or are using other investigational drug or are within 5 half-lives after the last dose of the investigational drug.
13. Used a subunit or inactivated vaccine within 14 days or an attenuated live vaccine within 1 month (30 days) before the study vaccination, or plan to receive any other vaccines except for the seasonal influenza vaccine, or other vaccines for emergency use (e.g., to prevent tetanus and rabies) during the study.
14. Prior receipt of any investigational or licensed COVID-19 vaccine except for the primary vaccination with inactivated vaccines according to the protocol, or plan to receive any COVID-19 vaccine except for the investigational products during the study stage.
15. Suspected or known current alcohol or drug dependency.
16. Having contraindications for intramuscular injection or intravenous blood sampling.
17. Pregnancy, lactation or plan to become pregnant within 90 days after receiving study vaccine.
18. Staff of study site, sponsor, and contract research organization (CRO) taking part in study conduct.
19. At investigator's discretion, any other significant disease, disorder or finding that may increase the risk because of participation in the study, or prevent from participation in the study, or impair interpretation of the study data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Immunogenicity at Phase II Study | at 14 days after the booster vaccination
  The GMT of live-virus neutralizing antibody against SARS-CoV-2 prototype at 14 days after the booster vaccination.
Immunogenicity at Phase II Study | at14 days after the booster vaccination
  The SCR of live-virus neutralizing antibody against SARS-CoV-2 prototype at 14 days after the booster vaccination
Safety at Phase II Study | within 7 days after the booster vaccination
  The occurrence of solicited local and systemic adverse events (AEs) within 7 days after the booster vaccination
Safety at Phase II Study | within 28 days after the booster vaccination
  The occurrence of unsolicited AEs within 28 days after the booster vaccination
Safety at Phase II Study | till 6 months after the booster vaccination
  The occurrence of serious adverse events (SAEs) and adverse events of special interest (AESIs) till 6 months after the booster vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Suad Al Hannawi, Dr., Principal Investigator — AI Kuwait Hospital
Locations (1):
- AI Kuwait Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available

REFERENCES:
- [Derived] Balgos A, Hannawi S, Chen WL, Abuquta A, Safeldin L, Hassan A, Alamadi A, Tirador L, Jaen AM, Villalobos RE, Mo C, Yue ZJ, Ma Y, Wang QS, Wen RD, Yao Z, Yu JP, Yao WR, Zhang JH, Hong KX, Liu Y, Li JX. Immunogenicity and safety of boosting with a recombinant two-component SARS-CoV-2 vaccine: two randomized, parallel-controlled, phase 2 studies. Expert Rev Vaccines. 2024 Jan-Dec;23(1):419-431. doi: 10.1080/14760584.2024.2334423. Epub 2024 Apr 2. PMID 38529685